CLINICAL TRIAL: NCT06384638
Title: Efficacy of Locally Delivered Coconut Oil in Management of Stage II and III Grade B Periodontitis. A Randomized Controlled Clinical Trial
Brief Title: Coconut Oil in Treatment of Periodontitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Radwa Elsherif, lecturer of oral medicine, periodontology and oral diagnosis at Misr University for science and technology, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: coconut periodontitis
Record Dates: First submitted 2024-04-19; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Diseases
Keywords: Periodontitis; coconut oil; scaling and debridement
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Tooth Exfoliation; Debridement

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Active Comparator): coconut oil as topical application as adjunctive to scaling and root debridement
  Interventions: Biological: topical application of coconut oil; Other: scaling and debridement
- control (Active Comparator): scaling and root debridement
  Interventions: Other: scaling and debridement

INTERVENTIONS:
Biological: topical application of coconut oil — topical application of coconut oil
  Arms: interventional
Other: scaling and debridement — scaling and debridement

SUMMARY:
Virgin Coconut Oil (VCO) is a vegetable oil extracted from coconut fleshcontains unsaturated fatty acids in the form of oleic acid and linoleic acid and flavonoids which function as anti-inflammatory. Periodontitis is an inflammatory disease of the periodontal tissues with a high prevalence worldwide. The main etiology of plaque periodontitis is biofilm containing colonies of pathogenic microorganisms. The aim of the study is to evaluate and compare the effect of scaling and root debridement alone versus the use of topically applied coconut oil as adjunctive to scaling and root debridement in treatment of Stage II and III Grade B periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* patients age group >35 years without ant systemic disease
* Willing to take part in the study. Patients with more than 16 natural teeth and have test teeth with both mesial and distal neighboring teeth with periodontitis with clinical attachment loss >3 mm and radiographic percentage of bone loss/age ranged between 0.25 to 1.
* Patients with no history of allergies to coconut

Exclusion Criteria:

* smokers
* pregnant
* lactating women
* Teeth with both endodontic-periodontal lesion.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
clinical parameters | 3 months
  clinical attachment loss
clinical parameters | 3 months
  Probing depth

SECONDARY OUTCOMES:
Biological parameters | 3 months
  Tumor necrosis factor alpha (TNF- α) levels by using ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry at MUST, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No